CLINICAL TRIAL: NCT05902936
Title: Short Term Clinical and Radiographic Evaluation of Nano Bioactive Glass Combined With i-PRF Scaffold in Vital Pulp Treatments in Mature Permanent Mandibular Molars: A Triple Blinded "Randomized Controlled Trial"
Brief Title: Evaluation of Nano Bioactive Glass Combined With i-PRF Scaffold in Vital Pulp Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Peter Nabil Naguib, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO3-7-2
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pulpitis - Irreversible; Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * The participant will be blinded to the materials will be used during the pulpotomy process.
  * The outcome assessors will be blinded.
  * The operator will not be blinded for both materials during pulpotomy procedure as the two materials having different colors and different handling techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): After control of bleeding in teeth allocated to the control group i-PRF is to be injected first. The i-PRF will be injected into the root canal to a level 3 mm below the cementoenamel junction (CEJ) then a layer of premixed bioceramic putty is to be added for coronal sealing.
  Interventions: Procedure: Pulpotomy for mature permanent mandibular molars
- Intervention group (Active Comparator): After control of bleeding in teeth allocated to the intervention group, i-PRF is to be mixed with Nano bioactive glass (Nano-BAG) powder to a putty consistency and injected into the root canal to a level 3 mm below the cementoenamel junction (CEJ), then a layer of premixed bioceramic putty is to be added for coronal sealing.
  Interventions: Procedure: Pulpotomy for mature permanent mandibular molars

INTERVENTIONS:
Procedure: Pulpotomy for mature permanent mandibular molars — Performing pulpotomy for mature teeth that involves removal of the coronal pulp tissue that is diseased or inflammed followed by placement of a biocompatible material with the intent of maintaining the vitality of the remaining radicular pulp tissue.
  Other Names: Vital pulp therapy

SUMMARY:
With consideration of the previous studies regarding the properties of i-PRF, it will be used in combination with another bioactive material: (Nano-BAG) versus using of i-PRF only as a pulpotomy material with using a premixed bioceramic putty as a coronal sealing material in both cases, to evaluate if there is a difference in the success rate of pulpotomy in case of using Nano-BAG in combination with i-PRF

So, in this study the investigators will use Nano-BAG in combination with i-PRF as a material for pulpotomy in cases of mature permanent mandibular molars and compare its outcomes with using i-PRF only and in both cases pulpotomy material will be covered with a layer of premixed bioceramic putty for coronal sealing.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the outcome of i-PRF mixed with Nano-bioactive Glass powder and i-PRF alone covered with a layer of premixed bioceramic putty when used as a material for pulpotomy in terms of relieving pain and maintaining the radicular pulp vitality and inducing dentin bridge formation in mature permanent mandibular molars.

Research Question:

Will i-PRF mixed with Nano-BAG and covered with premixed bioceramic putty gives similar results in relieving pain , conservation of the radicular pulp vitality and dentin bridge formation compared with i-PRF alone covered with premixed bioceramic putty when using it as a material for pulpotomy in mature permanent mandibular molars?

Interventions:

A- Intervention for each group

a- General operative procedures

• Eligible patients will be randomized in equal proportions between the two groups.

Patients of the two groups will be subjected to:

* Diagnosis using diagnostic chart (appendix A) and selected according to inclusion and exclusion criteria
* Comprehensive clinical examination and understanding of patients' chief complaint and needs.
* Standard preoperative digital x-ray for all patients.

B- Intra operative procedures: (For both groups) Before anesthesia, surfaces of the teeth will be cleaned to be free of debris, calculus and plaque. Teeth will first be dried and isolated with cotton rolls and a tooth paste will be applied on the buccal face of the crown as an interface media. An electric pulp tester (EPT) probe will be placed on the sound coronal third of the labial surface and the responses will be recorded before starting the treatment. The contra lateral tooth will be tested first for comparison and then the subjected tooth will be checked.

The procedures will be performed under local anesthesia with Lidocaine 2% and adrenaline 1/100,000. Teeth will be isolated with rubber dam.

All carious tissue and old restoration (if present) will be removed with a diamond stone size 1 in a high speed hand piece with coolant , once the pulp is exposed the diamond stone will be changed and another sterile one will be used for complete deroofing of the pulp chamber. Then a sharp sterile excavator will be used for amputation of the coronal pulp tissue to the level of the root canal orifices.

Haemostasis will be achieved by pressing sterile cotton pellets soaked with sterile saline and damped into the cavity for 5-10 minutes over the pulp stumps (If haemostasis cannot be achieved after 10 mins, the tooth should undergo root canal treatment)

Care should be taken to minimize the time elapsed between coronal pulp amputation and placement of pulpotomy agent. The teeth will be then divided into two groups depending on the pulpotomy agents. I-PRF will be prepared according to Choukroun's technique by drawing a whole blood sample from the median cubital vein into a 10 ml plain test tubes (Non-citrated) to prevent blood coagulation then it will be centrifuged immediately using a table top centrifuge at 700 rpm for 3 mins The whole blood sample that will be obtained consists of three layers: the top most layer of acellular platelet poor plasma, the middle layer of platelet rich fibrin, and the bottom most layer of red blood corpuscles. The upper yellow fluid liquid (i-PRF) will be collected as close as possible to the layer of red blood cell.

Group A (the control group) :

After control of bleeding in teeth allocated to the control group i-PRF is to be injected first. The i-PRF will be injected into the root canal to a level 3 mm below the cementoenamel junction (CEJ).

Group B (In the intervention group):

After control of bleeding in teeth allocated to the intervention group, i-PRF is to be mixed with Nano-BAG powder to a putty consistency and injected into the root canal to a level 3 mm below the cementoenamel junction (CEJ), then a layer of premixed bioceramic putty is to be added for coronal sealing.

Coronal Sealing:

After a period of 10-15-minutes is allowed for coagulation, the coronal sealing material will be applied. The premixed bioceramic putty is dispensed on a sterile glass slab using a flat sided sterile plastic instrument. The material is applied over the coagulated scaffold in both groups using a dedicated carrier (MAP one) The material is adapted over the scaffold using light pressure adaptation with a sterile micro-brush of suitable size.

Final restoration:

A thin layer of resin-modified glass ionomer cement (RMGIC) to be applied directly over the coronal seal. Composite Resin material is to be used as a final restoration.

ELIGIBILITY:
Inclusion Criteria:

* • Patients suffering from symptomatic irreversible pulpitis.

  * Tooth should give positive response to cold test
  * Heamostatis should be achieved after complete pulpotomy
  * Diagnosis is irreversible pulpitis with/without apical periodontitis
  * The tooth is restorable and free from advanced periodontal disease
  * Tooth is free from cracks or splits
  * Patients should be free from any systemic disease that may affect normal healing and predictable outcomes.
  * Patients who will agree to the consent and will commit to follow-up period.
  * Patients with mature root (closed apices)
  * Teeth with no periapical lesion, resorption or widening.
  * Soft tissues around the tooth are normal with no swelling or sinus tract
  * Mandibular posterior teeth only will be involved.

Exclusion Criteria:

* • Patients with immature root apices.

  * Patients with any systemic disease that may affect normal healing.
  * Patients with periapical lesions or infections.
  * If heamostasis couldn't be achieved within 5-10 minutes
  * Pregnant females.
  * Patients who could/would not participate in a 6 months follow-up.
  * Patients with fistula or swelling
  * Patients with necrotic pulp.
  * Patients with old age.
  * Badly destructed teeth
  * Teeth that are non-restorable
  * Teeth that require post and core build up

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Pain measurement (change is being assessed) | After 24 hours and up to 7 days for postoperative pain evaluation using Visual Analogue Scale.
  Measurement of the change in pain intensity using Visual Analogue Scale from 0 to 10 where higher scores mean higher pain intensity

SECONDARY OUTCOMES:
Radiographic assesment (change is being assessed) | at 1 month , 3 months and 6 months
  Radiographic assesment of dentin bridge formation whether it is present or absent
Tooth sensibility (change is being assessed) | at 1 month , 3 months and 6 months
  Tooth sensibility will be assessed using Thermal (cold) test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No